CLINICAL TRIAL: NCT05100485
Title: A Novel Algorithm to Stratify Clinical Decompensation Risk in Patients With Compensated Advanced Chronic Liver Disease (CHESS2108)
Brief Title: Algorithm to Stratify Clinical Decompensation Risk in Patients With Compensated Advanced Chronic Liver Disease (CHESS2108)
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: Tianjin Second People's Hospital (Other); The Third People's Hospital of Taiyuan (Other); Ehime University Graduate School of Medicine (Other); Korea University Ansan Hospital (Other); Hyogo Medical University (Other); Zagazing University Faculty of Medicine (Unknown); Institute of Liver and Biliary Sciences (ILBS) (Unknown); Changi General Hospital (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Prof., Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS2108
Record Dates: First submitted 2021-10-20; First posted 2021-10-29 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Compensated Advanced Chronic Liver Disease
Keywords: liver stiffness; platelets; portal hypertension; varices; compensated advanced chronic liver disease
MeSH Terms: conditions — Hypertension, Portal; Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training cohort: Training cohort was used to developement the new algorithm for predicting liver decompensation.
  Interventions: Diagnostic Test: Esophagogasrtoduodendoscopy
- Validation cohort: Validation cohort was used to test the performance of the new algorithm in predicting liver decompensation.
  Interventions: Diagnostic Test: Esophagogasrtoduodendoscopy
- HVPG cohort: HVPG cohort, a cross-section cohort was used to study the diagnostic value of novel score for clinically significant portal hypertension.
  Interventions: Diagnostic Test: Esophagogasrtoduodendoscopy; Diagnostic Test: Hepatic venous pressure gradient

INTERVENTIONS:
Diagnostic Test: Esophagogasrtoduodendoscopy — Esophagogasrtoduodendoscopy was used to detech the presence of varices.
Diagnostic Test: Hepatic venous pressure gradient — A method used to eveluate the portal pressure
  Groups: HVPG cohort

SUMMARY:
Compensated advanced chronic liver disease (cACLD) commonly indicates severe fibrosis and compensated cirrhosis at risk of developing clinically significant portal hypertension (CSPH) and hepatic decompensation. The presence of CSPH (defined as hepatic venous pressure gradient [HVPG] ≥ 10 mmHg) is the strongest predictor of hepatic decompensation. However, HVPG measurement is invasive, operator dependent, and not widely available. According to the 2021 updated EASL Clinical Practice Guidelines, cACLD patients who did not meet the Baveno VI criteria but had any of the two variables (LSM > 20 kPa or PLT < 150 × 109/L) were suggested to perform screening endoscopy and HVPG measurement. However, the number of cACLD patients with unfavorable Baveno VI status is huge, no detailed risk stratifications existed at this timepoint. This study intended to investigate a novel algorithm to stratify the decompensation risk in patients with cACLD.

DETAILED DESCRIPTION:
Compensated advanced chronic liver disease (cACLD) commonly indicates severe fibrosis and compensated cirrhosis at risk of developing clinically significant portal hypertension (CSPH) and hepatic decompensation. The presence of CSPH (defined as hepatic venous pressure gradient [HVPG] ≥ 10 mmHg) is the strongest predictor of hepatic decompensation. However, HVPG measurement is invasive, operator dependent, and not widely available. According to the 2021 updated EASL Clinical Practice Guidelines, cACLD patients who did not meet the Baveno VI criteria but had any of the two variables (LSM > 20 kPa or PLT < 150 × 109/L) were suggested to perform screening endoscopy and HVPG measurement. However, the number of cACLD patients with unfavorable Baveno VI status is huge, no detailed risk stratifications existed at this timepoint. This international multicenter cohort study intended to investigate a novel algorithm to stratify the decompensation risk in patients with cACLD.

ELIGIBILITY:
Training and Validation cohort

Inclusion Criteria:

1. age above or equal to 18-year-old,
2. fulfilled diagnosis of cACLD based on radiological, histological features of severe fibrosis or cirrhosis according to the Baveno VI consensus.

Exclusion Criteria:

1. prior hepatic decompensation,
2. hepatocellular carcinoma,
3. prior liver transplantation,
4. portal vein thrombosis,
5. antiplatelet or anticoagulation,
6. without screening endoscopy within six months of transient elastography,
7. alcoholic cirrhosis with significant ongoing alcohol intake,
8. presence of gastric varix,
9. incomplete follow-up data.

HVPG cohort.

Inclusion Criteria:

1. age above or equal to 18-year-old,
2. fulfilled diagnosis of cACLD based on radiological, histological features of severe fibrosis or cirrhosis according to the Baveno VI consensus.

Exclusion Criteria:

1. prior hepatic decompensation,
2. hepatocellular carcinoma,
3. prior liver transplantation,
4. portal vein thrombosis,
5. antiplatelet or anticoagulation,
6. without screening endoscopy within six months of transient elastography,
7. alcoholic cirrhosis with significant ongoing alcohol intake,
8. presence of gastric varix,
9. non-sinusoidal portal hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an international, multicenter cohort study initialed by Portal Hypertension Alliance in China (CHESS) and eligible patients will enroll from China, Japan, Southern Korea, Egypt, Singapore, and India.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of a novel algorithm for predicting liver decompensation. | 3 years
  Aims to investigate the accuracy of the novel algorithm to stratify decompensation risk in patients with cACLD.

SECONDARY OUTCOMES:
The accuracy of the novel alogrithm for predicting clinically significant portal hypertension. | 1 years
  HVPG cohort was used to evaluate the accuracy of the novel alogrithm for predicting clinically significant portal hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, MD, Study Chair — Lanzhou University First Affiliated Hospital; Qing Xie, MD, Principal Investigator — Shanghai Jiao Tong university affiliated Ruijin Hospital; Jia Li, MD, Principal Investigator — Tianjin Second People's Hospital; Yu Jun Wong, MD, Principal Investigator — Changi General Hospital; Masashi Hirooka, MD, Principal Investigator — Ehime University Graduate School of Medicine; Hirayuki Enomoto, MD, Principal Investigator — Hyogo Medical University; Tae Hyung Kim, MD, Principal Investigator — Korea UniversityAnsan Hospital; Amr Shaaban Hanafy, MD, Principal Investigator — Zagazig University; Ying Guo, MD, Principal Investigator — The Third People's Hospital of Taiyuan; Shiv Sarin, MD, Principal Investigator — Institute of Liver and Biliary Sciences (ILBS)
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Villanueva C, Albillos A, Genesca J, Garcia-Pagan JC, Calleja JL, Aracil C, Banares R, Morillas RM, Poca M, Penas B, Augustin S, Abraldes JG, Alvarado E, Torres F, Bosch J. beta blockers to prevent decompensation of cirrhosis in patients with clinically significant portal hypertension (PREDESCI): a randomised, double-blind, placebo-controlled, multicentre trial. Lancet. 2019 Apr 20;393(10181):1597-1608. doi: 10.1016/S0140-6736(18)31875-0. Epub 2019 Mar 22. PMID 30910320
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines on non-invasive tests for evaluation of liver disease severity and prognosis - 2021 update. J Hepatol. 2021 Sep;75(3):659-689. doi: 10.1016/j.jhep.2021.05.025. Epub 2021 Jun 21. PMID 34166721
- [Background] Albilllos A, Garcia-Tsao G. Classification of cirrhosis: the clinical use of HVPG measurements. Dis Markers. 2011;31(3):121-8. doi: 10.3233/DMA-2011-0834. PMID 22045397
- [Background] Ripoll C, Groszmann R, Garcia-Tsao G, Grace N, Burroughs A, Planas R, Escorsell A, Garcia-Pagan JC, Makuch R, Patch D, Matloff DS, Bosch J; Portal Hypertension Collaborative Group. Hepatic venous pressure gradient predicts clinical decompensation in patients with compensated cirrhosis. Gastroenterology. 2007 Aug;133(2):481-8. doi: 10.1053/j.gastro.2007.05.024. Epub 2007 May 21. PMID 17681169
- [Background] Bosch J, Abraldes JG, Berzigotti A, Garcia-Pagan JC. The clinical use of HVPG measurements in chronic liver disease. Nat Rev Gastroenterol Hepatol. 2009 Oct;6(10):573-82. doi: 10.1038/nrgastro.2009.149. Epub 2009 Sep 1. PMID 19724251
- [Background] Thabut D, Bureau C, Layese R, Bourcier V, Hammouche M, Cagnot C, Marcellin P, Guyader D, Pol S, Larrey D, De Ledinghen V, Ouzan D, Zoulim F, Roulot D, Tran A, Bronowicki JP, Zarski JP, Goria O, Cales P, Peron JM, Alric L, Bourliere M, Mathurin P, Blanc JF, Abergel A, Serfaty L, Mallat A, Grange JD, Attali P, Bacq Y, Wartelle-Bladou C, Dao T, Pilette C, Silvain C, Christidis C, Capron D, Bernard-Chabert B, Hillaire S, Di Martino V, Sutton A, Audureau E, Roudot-Thoraval F, Nahon P; ANRS CO12 CirVir group. Validation of Baveno VI Criteria for Screening and Surveillance of Esophageal Varices in Patients With Compensated Cirrhosis and a Sustained Response to Antiviral Therapy. Gastroenterology. 2019 Mar;156(4):997-1009.e5. doi: 10.1053/j.gastro.2018.11.053. Epub 2019 Feb 13. PMID 30768988
- [Background] Abraldes JG, Bureau C, Stefanescu H, Augustin S, Ney M, Blasco H, Procopet B, Bosch J, Genesca J, Berzigotti A; Anticipate Investigators. Noninvasive tools and risk of clinically significant portal hypertension and varices in compensated cirrhosis: The "Anticipate" study. Hepatology. 2016 Dec;64(6):2173-2184. doi: 10.1002/hep.28824. Epub 2016 Oct 27. PMID 27639071
- [Background] Chen RC, Cai YJ, Wu JM, Wang XD, Song M, Wang YQ, Zheng MH, Chen YP, Lin Z, Shi KQ. Usefulness of albumin-bilirubin grade for evaluation of long-term prognosis for hepatitis B-related cirrhosis. J Viral Hepat. 2017 Mar;24(3):238-245. doi: 10.1111/jvh.12638. Epub 2016 Nov 14. PMID 27862671